CLINICAL TRIAL: NCT03725852
Title: A Phase II Randomized, Double-blind, Placebo-controlled, 26-week Study to Evaluate the Efficacy, Safety and Tolerability of GLPG1205 in Subjects With Idiopathic Pulmonary Fibrosis
Brief Title: A Clinical Study to Test How Effective and Safe GLPG1205 is for Participants With Idiopathic Pulmonary Fibrosis (IPF)
Acronym: PINTA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG1205-CL-220; 2017-004302-18 (EudraCT Number)
Record Dates: First submitted 2018-06-08; First posted 2018-10-31 (Actual); Results first posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-08

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — GLPG1205

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GLPG1205 100 mg (Experimental): Participants will receive GLPG1205 100 milligrams (mg) (2 capsules x 50 mg), orally once daily for 26 weeks in addition to the local standard of care. Standard of care includes nintedanib, pirfenidone, or neither nintedanib nor pirfenidone.
  Interventions: Drug: GLPG1205
- Placebo (Placebo Comparator): Participants will receive GLPG1205 matching placebo, orally once daily (as 2 capsules) for 26 weeks in addition to the local standard of care. Standard of care includes nintedanib, pirfenidone, or neither nintedanib nor pirfenidone.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLPG1205 — GLPG1205 will be provided as an oral hard gelatin capsule.
  Arms: GLPG1205 100 mg
Drug: Placebo — GLPG1205 matching placebo will be provided as an oral hard gelatin capsule.
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, parallel-group, placebo-controlled, multicenter, exploratory Phase 2 study including participants with Idiopathic Pulmonary Fibrosis (IPF), investigating GLPG1205 in addition to the local standard of care (defined as receiving nintedanib, pirfenidone, or neither nintedanib nor pirfenidone).

ELIGIBILITY:
Inclusion criteria:

Participants who meet all of the following criteria are eligible for the study:

* A diagnosis of IPF within 5 years prior to the screening visit as per applicable American Thoracic Society (ATS)/European Respiratory Society(ERS)/Japanese Respiratory Society (JRS)/Latin American Thoracic Association (ALAT) guideline. Participants receiving local standard of care for the treatment of IPF, defined as either pirfenidone or nintedanib at a stable dose for at least 8 weeks before screening, and during screening; or neither pirfenidone nor nintedanib (for any reason). A stable dose is defined as the highest tolerated dose. Prednisone at steady dose less than or equal to 10 mg/day or equivalent glucocorticoid dose is allowed (stabilized 4 weeks prior to screening and continued without variation of dose or regimen). Supportive care like supplemental oxygen or pulmonary rehabilitation is allowed.
* Meeting all of the following criteria at screening and during the screening period:

  * Forced vital capacity (FVC) greater than or equal to 50% predicted of normal
  * Disease progression, defined as a decline of FVC (% predicted or milliliters [mL]) at the investigator's discretion, during the 9 months prior to the screening period and confirmed at the screening visit
  * Diffusing capacity for the lungs for carbon monoxide (DLCO) greater than or equal to 30% predicted of normal (corrected for hemoglobin)
  * Ratio of forced expiratory volume in one second (FEV1) to FVC greater than or equal to 0.70
* In a stable condition and suitable for study participation based on the results of a medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), and laboratory evaluation. Stable condition is based on the clinical judgment of the investigator, co-morbidities should be treated according to the local applicable guidelines. Concomitant medication for chronic comorbidities should be stabilized from 4 weeks before screening and during the screening period (stable defined as no clinically relevant change according to the investigator's judgement).
* Able to walk at least 150 meters during the 6 Minute Walk Test (6MWT) at screening; without having a contraindication to perform the 6MWT.

This list only describes the key inclusion criteria.

Exclusion criteria:

Participants meeting one or more of the following criteria cannot be selected for this study:

* Known hypersensitivity to any of the investigational medicinal product (IMP) ingredients or a history of a significant allergic reaction to any drug as determined by the investigator (e.g. anaphylaxis requiring hospitalization).
* Current immunosuppressive condition (e.g. human immunodeficiency virus [HIV] infection, congenital, acquired, medication induced, organ transplantation).
* Positive blood testing for hepatitis B surface antigen (HBS Ag) or hepatitis C virus (HCV) antibody (if positive, confirmed by HCV ribonucleic acid [RNA] positivity). Note: Participants with a resolved hepatitis A at least 3 months prior to first dosing of the IMP can be included.
* History of malignancy within the past 5 years (except for carcinoma in situ of the uterine cervix, basal cell carcinoma of the skin that has been treated with no evidence of recurrence, and prostate cancer medically managed through active surveillance or watchful waiting, and squamous cell carcinoma of the skin if fully resected).
* Acute IPF exacerbation within 3 months prior to screening and during the screening period.
* Lower respiratory tract infection requiring antibiotics within 4 weeks prior to screening and/or during the screening period.
* Interstitial lung disease associated with known primary diseases (e.g. sarcoidosis, amyloidosis), exposures (e.g. radiation, silica, asbestos, coal dust), and drugs (e.g. amiodarone).
* History of lung volume reduction surgery or lung transplant.
* Unstable cardiovascular, pulmonary (other than IPF) or other disease within 6 months prior to screening or during the screening period (e.g. coronary heart disease, heart failure, stroke).
* Participant participating in a drug, device or biologic investigational research study, concurrently with the current study, within 12 weeks or 5-half-lives of the agent, whichever is longer, prior to screening, or prior participation in an investigational drug antibody/biologic study within 6 months prior to screening.

This list only describes the key exclusion criteria.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2020-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Seemayer, MD, Study Director — Galapagos NV
Locations (36):
- Bulgaria (3):
  - Specialized Hospital for Active Treatment Pleven, Pleven
  - SHATPPD Dr. Dimitar Gramatikov, Ruse Ltd., Rousse
  - Acibadem City Clinic Tokuda Hospital, EAD, Sofia
- Croatia (3):
  - Klinicki Bolnicki Centar Rijeka - Susak, Rijeka
  - Klinička Bolnica Dubrava, Zagreb
  - Klinički Bolnički Centar Zagreb - Klinika Za Plućne Bolesti Jordanovac, Zagreb
- Finland (2):
  - Helsinki University Hospital Heart and Lung Center, Helsinki
  - Tampere University Hospital, Tampere
- France (10):
  - Hôpital Avicenne, Bobigny
  - CHU de Brest - Hôpital Cavale Blanche, Brest
  - CHU de Lyon - Hôpital Louis Pradel, Bron
  - CHU de Grenoble, La Tronche
  - Hôpital Albert Calmette, Lille
  - CHU de Nice - Hôpital Pasteur, Nice
  - Hôpital Européen Georges Pompidou (HEGP), Paris
  - Hôpital Larrey, Toulouse
  - CHRU de Tours - Hôpital Bretonneau, Tours
  - Hôpitaux Prives de Metz (HPMetz) - Hôpital Robert Schuman, Vantoux
- National Oncology Centre - The Royal Hospital Muscat, Muscat, Oman
- Romania (4):
  - Institutul de Pneumoftiziologie Marius Nasta, Bucharest
  - Spitalul Clinic De Pneumoftiziologie Leon Daniello Cluj-Napoca, Cluj-Napoca
  - Spitalul Clinic de Pneumoftiziologie Iasi, Iași
  - Clinica Medicala Lavinia Davidescu, Oradea
- Slovakia (3):
  - ZAPA JJ s.r.o., Levice
  - Pľúcna Ambulancia Hrebenár, s.r.o., Spišská Nová Ves
  - National Institute of Tuberculosis, Pulmonary Diseases and Chest Surgery, Vyšné Hágy
- Sweden (3):
  - Universitetssjukhuset i Lund, Lund
  - Karolinska Universitetssjukhuset, Stockholm
  - Akademiska Sjukhuset - Uppsala Centrum for Cystisk Fibros, Uppsala
- Ukraine (7):
  - Dnipropetrovsk State Medical Academy - Dnipropetrovsk City Clinical Hospital No. 6, Dnipropetrovsk
  - The Ivano-Frankivsk National Medical Univeristy, Ivano-Frankivsk
  - Communal Nonprofit Enterprise City Clinical Hospital, Kharkiv
  - Municipal Institution "Kherson city clinical hospital named after E.E. Karabelesh", Kherson
  - National Institute of Phthisiology and Pulmonology named after F.G. Yanovskyi of NAMS of Ukraine, Kyiv
  - Odessa Regional Hospital, Odesa
  - Vinnitsa Regional Clinical Hospital im. N.I. Pirogov, Vinnytsia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Strambu IR, Fagard L, Ford P, Van Der Aa T, De Haas-Amatsaleh A, Santermans E, Seemayer C. (2020). Idiopathic pulmonary fibrosis (IPF): observations from a Phase 2 trial of GLPG1205 (PINTA). Abstract for European Respiratory Society International Congress 7-9 September 2020.
- [Derived] Strambu IR, Seemayer CA, Fagard LMA, Ford PA, Van der Aa TAK, de Haas-Amatsaleh AA, Modgill V, Santermans E, Sondag EN, Helmer EG, Maher TM, Costabel U, Cottin V. GLPG1205 for idiopathic pulmonary fibrosis: a phase 2 randomised placebo-controlled trial. Eur Respir J. 2023 Mar 2;61(3):2201794. doi: 10.1183/13993003.01794-2022. Print 2023 Mar. PMID 36328358

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Bulgaria, Croatia, Finland, France, Oman, Romania, Slovakia, Sweden, and Ukraine. The first participant was screened on 27 Sep 2018. The last study visit occurred on 14 Aug 2020.
Pre-assignment Details: A total of 155 participants were screened, of which 86 participants were considered ineligible. Out of 69 enrolled participants, 1 participant met an exclusion criterion pre-dose and was therefore excluded.
Groups:
- GLPG1205 100 mg: Participants received GLPG1205 100 milligrams (mg) (2 capsules x 50 mg), orally once daily for 26 weeks in addition to the local standard of care. Standard of care included nintedanib, pirfenidone, or neither nintedanib nor pirfenidone.
- Placebo: Participants received GLPG1205 matching placebo, orally once daily (as 2 capsules) for 26 weeks in addition to the local standard of care. Standard of care included nintedanib, pirfenidone, or neither nintedanib nor pirfenidone.
Period: Overall Study
Arm/Group | GLPG1205 100 mg | Placebo
Started | 45 | 23
Completed | 41 | 23
Not Completed | 4 | 0
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Travel restrictions due to COVID-19 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) consisted of all randomized participants who received at least 1 dose of study drug.
Groups:
- GLPG1205 100 mg: Participants received GLPG1205 100 mg (2 capsules x 50 mg), orally once daily for 26 weeks in addition to the local standard of care. Standard of care included nintedanib, pirfenidone, or neither nintedanib nor pirfenidone.
- Total: Total of all reporting groups
Arm/Group | GLPG1205 100 mg | Placebo | Total
Number analyzed (Participants) | 45 | 23 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.5 (6.8) | 68.3 (5.5) | 69.8 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 18
  Male | 33 | 17 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 45 | 23 | 68
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 32 | 17 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 6 | 17

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Forced Vital Capacity (FVC) at Week 26
Description: Forced vital capacity (FVC) (in milliliter [mL]) is the maximum amount of air exhaled from lungs by a participant after taking their deepest possible breath, as measured by spirometry.
Time Frame: Baseline, Week 26
Population: Participants in the full analysis set (FAS) (consisted of all randomized participants who received at least 1 dose of the study drug) with available data were analyzed.
Measure: Mean (Standard Error); unit: mL
Arm/Group | GLPG1205 100 mg | Placebo
Number analyzed (Participants) | 45 | 23
mL
  Baseline | 2865.43 (103.544) | 2817.08 (167.773)
  Change at Week 26: number analyzed (Participants) | 29 | 20
  Change at Week 26 | -31.29 (42.398) | -79.47 (32.838)
Statistical Analysis 1: Comparison: GLPG1205 100 mg vs Placebo; Change at Week 26; Test type: Superiority; p = 0.495, ANCOVA — P-value was based on an analysis of covariance (ANCOVA) model at each time point including treatment, sex, stratum (nintedanib, pirfenidone or neither), age, height, and baseline value as covariates; Least square (LS) mean difference = 42.33, 95% CI 2-sided [-81.84 to 166.49], Standard Error of Mean 61.483

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs, TEAEs Related to Study Drug, and TEAEs Leading to Study Drug Discontinuation
Description: An adverse event (AE) was any untoward medical occurrence in a participant administered study drug and which did not necessarily have a causal relationship with study drug. A TEAE was any AE with an onset date on or after the start of study drug intake and no later than 30 days after last dose of study drug, or any worsening of any AE on or after the start of study drug intake. A serious AE was defined as an AE that resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was medically significant.
Time Frame: First dose date up to 30 days after the last dose of study drug (maximum up to 263 days)
Population: Participants in the FAS population were analyzed.
Measure: Number; unit: participants
Arm/Group | GLPG1205 100 mg | Placebo
Number analyzed (Participants) | 45 | 23
participants
  TEAEs | 36 | 18
  Serious TEAEs | 9 | 1
  TEAEs related to study drug | 20 | 3
  TEAEs leading to study drug discontinuation | 10 | 0
Statistical Analysis 1: Comparison: GLPG1205 100 mg vs Placebo; TEAEs; Test type: Superiority; Difference in Percentage = 1.7, 95% CI 2-sided [-17.3 to 24.5] — 95% CI for difference calculated using the method of Miettinen and Nurminen
Statistical Analysis 2: Comparison: GLPG1205 100 mg vs Placebo; Serious TEAEs; Test type: Superiority; Difference in Percentage = 15.7, 95% CI 2-sided [-3.0 to 30.7] — 95% CI for difference calculated using the method of Miettinen and Nurminen
Statistical Analysis 3: Comparison: GLPG1205 100 mg vs Placebo; TEAEs related to study drug; Test type: Superiority; Difference in Percentage = 31.4, 95% CI 2-sided [8.2 to 49.4] — 95% CI for difference calculated using the method of Miettinen and Nurminen
Statistical Analysis 4: Comparison: GLPG1205 100 mg vs Placebo; TEAEs leading to study drug discontinuation; Test type: Superiority; Difference in Percentage = 22.2, 95% CI 2-sided [6.7 to 36.4] — 95% CI for difference calculated using the method of Miettinen and Nurminen

3. Secondary Outcome: Time to Any Major Events Depicted by Cumulative Percentage of Participants With All-cause Deaths, Respiratory-related Deaths, All-cause Hospitalizations, and Respiratory-related Hospitalizations
Description: Treatment effect on time to death (all-cause and respiratory-related)/hospitalization (all-cause and respiratory-related) were assessed using the log-rank test. Kaplan-Meier estimates were derived for the probability of death (all-cause and respiratory-related)/hospitalization (all-cause and respiratory-related). Cumulative percentage of participants with all-cause deaths, respiratory-related deaths, all-cause hospitalizations, and respiratory-related hospitalizations were reported.
Time Frame: Day 1 up to Week 30
Population: Participants in the FAS population were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GLPG1205 100 mg | Placebo
Number analyzed (Participants) | 45 | 23
percentage of participants
  All-cause deaths | 3.1 [0.4 to 20.2] | 0 [NA to NA] — Data could not be estimated as all participants in this group were censored.
  Respiratory-related deaths | 3.1 [0.4 to 20.2] | 0 [NA to NA] — Data could not be estimated as all participants in this group were censored.
  All-cause hospitalizations | 16.6 [8.3 to 31.9] | 4.3 [0.6 to 27.1]
  Respiratory-related hospitalizations | 2.8 [0.4 to 18.1] | 4.3 [0.6 to 27.1]
Statistical Analysis 1: Comparison: GLPG1205 100 mg vs Placebo; All-cause deaths; Test type: Superiority; p = 0.397, Log Rank
Statistical Analysis 2: Comparison: GLPG1205 100 mg vs Placebo; Respiratory-related deaths; Test type: Superiority; p = 0.397, Log Rank
Statistical Analysis 3: Comparison: GLPG1205 100 mg vs Placebo; All-cause hospitalizations; Test type: Superiority; p = 0.131, Log Rank
Statistical Analysis 4: Comparison: GLPG1205 100 mg vs Placebo; Respiratory-related hospitalizations; Test type: Superiority; p = 0.762, Log Rank

4. Secondary Outcome: Change From Baseline in Total Distance Walked in Six-minute Walk Test (6MWT) at Week 26
Description: The 6-MWT depicts the total distance covered by a participant during 6 minutes of walking.
Time Frame: Baseline, Week 26
Population: Participants in the FAS population with available data were analyzed.
Measure: Mean (Standard Error); unit: meters
Arm/Group | GLPG1205 100 mg | Placebo
Number analyzed (Participants) | 45 | 23
meters
  Baseline | 412.6 (18.53) | 391.8 (25.72)
  Change at Week 26: number analyzed (Participants) | 26 | 19
  Change at Week 26 | -16.6 (10.56) | -8.7 (10.43)
Statistical Analysis 1: Comparison: GLPG1205 100 mg vs Placebo; Change at Week 26; Test type: Superiority; p = 0.565, ANCOVA — P-value was based on an ANCOVA model at Week 26 including treatment, stratum (nintedanib, pirfenidone or neither) and baseline 6MWT distance as covariates; Weighted LS mean difference = -9.11, 95% CI 2-sided [-40.87 to 22.64], Standard Error of Mean 15.713

5. Secondary Outcome: Change From Baseline in St.George's Respiratory Questionnaire (SGRQ) Total Score at Week 26
Description: The SGRQ is a 50-item paper questionnaire designed to measure and quantify the impact of chronic respiratory disease on health-related quality of life (QOL) and well-being, split into 3 domains: symptoms (assessing the frequency and severity of respiratory symptoms), activity (assessing the effects of breathlessness on mobility and physical activity), and impact (assessing the psychosocial impact of the disease). Scores were weighted such that each domain score and the total score ranged from 0 to 100, with higher scores indicating the poorer health-related QOL.
Time Frame: Baseline, Week 26
Population: Participants in the FAS population with available data were analyzed.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | GLPG1205 100 mg | Placebo
Number analyzed (Participants) | 45 | 23
units on a scale
  Baseline | 45.363 (2.8518) | 48.599 (3.9497)
  Change at Week 26: number analyzed (Participants) | 29 | 19
  Change at Week 26 | -3.797 (2.6683) | -1.424 (2.7151)
Statistical Analysis 1: Comparison: GLPG1205 100 mg vs Placebo; Change at Week 26; Test type: Superiority; p = 0.673, ANCOVA — P-value was based on an ANCOVA model at Week 26 including treatment, stratum (nintedanib, pirfenidone or neither) and baseline SGRQ value as covariates; Weighted LS mean difference. = -1.58, 95% CI 2-sided [-9.06 to 5.91], Standard Error of Mean 3.710

6. Secondary Outcome: Change From Baseline in SGRQ Domain Score at Week 26
Description: The SGRQ is a 50-item paper questionnaire designed to measure and quantify the impact of chronic respiratory disease on health-related QOL and well-being, split into 3 domains: symptoms (assessing the frequency and severity of respiratory symptoms), activity (assessing the effects of breathlessness on mobility and physical activity), and impact (assessing the psychosocial impact of the disease). Scores were weighted such that each domain score ranged from 0 to 100, with higher scores indicating the poorer health-related QOL.
Time Frame: Baseline, Week 26
Population: Participants in the FAS population with available data were analyzed.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | GLPG1205 100 mg | Placebo
Number analyzed (Participants) | 45 | 23
units on a scale
  Baseline (symptoms score) | 49.454 (3.7439) | 56.059 (4.3333)
  Change at Week 26 (symptoms score): number analyzed (Participants) | 29 | 19
  Change at Week 26 (symptoms score) | -3.135 (2.6281) | -3.437 (4.4017)
  Baseline (activity score) | 58.243 (3.0224) | 59.454 (4.6140)
  Change at Week 26 (activity score): number analyzed (Participants) | 29 | 20
  Change at Week 26 (activity score) | -4.387 (3.5367) | 1.156 (3.6228)
  Baseline (impacts score) | 36.409 (3.1765) | 40.064 (4.2897)
  Change at Week 26 (impacts score): number analyzed (Participants) | 29 | 20
  Change at Week 26 (impacts score) | -3.460 (3.1330) | -1.412 (3.2971)
Statistical Analysis 1: Comparison: GLPG1205 100 mg vs Placebo; Change at Week 26: Symptoms score; Test type: Superiority; p = 0.875, ANCOVA — [p-value comment as in outcome 5, analysis 1]; Weighted LS mean difference = -0.72, 95% CI 2-sided [-9.98 to 8.53], Standard Error of Mean 4.591
Statistical Analysis 2: Comparison: GLPG1205 100 mg vs Placebo; Change at Week 26: Activity score; Test type: Superiority; p = 0.416, ANCOVA — [p-value comment as in outcome 5, analysis 1]; Weighted LS mean difference = -4.14, 95% CI 2-sided [-14.29 to 6.02], Standard Error of Mean 5.038
Statistical Analysis 3: Comparison: GLPG1205 100 mg vs Placebo; Change at Week 26: Impacts score; Test type: Superiority; p = 0.961, ANCOVA — [p-value comment as in outcome 5, analysis 1]; Weighted LS mean difference = -0.20, 95% CI 2-sided [-8.32 to 7.92], Standard Error of Mean 4.029

7. Secondary Outcome: Percentage of SGRQ Responders
Description: The SGRQ is a 50-item paper questionnaire designed to measure and quantify the impact of chronic respiratory disease on health-related QOL and well-being, split into 3 domains: symptoms (assessing the frequency and severity of respiratory symptoms), activity (assessing the effects of breathlessness on mobility and physical activity), and impact (assessing the psychosocial impact of the disease). Scores were weighted such that each domain score and total score ranged from 0 to 100, with higher scores indicating the poorer health-related QOL. SGRQ responders are those with absolute change from baseline in SGRQ total score less than or equal to -4 percent (%) at least once.
Time Frame: Baseline up to Week 26
Population: Participants in the FAS population with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | GLPG1205 100 mg | Placebo
Number analyzed (Participants) | 40 | 22
percentage of participants | 40.0 | 40.9
Statistical Analysis 1: Comparison: GLPG1205 100 mg vs Placebo; Test type: Superiority; p = 1.000, Fisher Exact

8. Secondary Outcome: Pre-dose Plasma Concentration (Ctrough) of GLPG1205 at Week 26
Description: GLPG1205 pre-dose plasma concentration (Ctrough) at Week 26 was reported applying the exclusion rules (e.g. dose reduction, discontinuation, samples flagged).
Time Frame: Week 26 (pre-dose)
Population: Participants in the pharmacokinetic (PK) analysis set (a subset of the FAS, including all participants who had available and evaluable plasma concentration data, excluding all protocol deviations or AEs that may have had an impact on the PK analysis) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | GLPG1205 100 mg
Number analyzed (Participants) | 25
nanograms per milliliter (ng/mL) | 4979.9 (2279.5)

9. Secondary Outcome: Pre-dose Plasma Concentration (Ctrough) of Nintedanib at Week 20
Description: Nintedanib pre-dose plasma concentration (Ctrough) at Week 20 was reported applying the exclusion rules (e.g. dose reduction, discontinuation, samples flagged).
Time Frame: Week 20 (pre-dose)
Population: Participants in the PK analysis set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | GLPG1205 100 mg | Placebo
Number analyzed (Participants) | 4 | 4
ng/mL | 14.58 (6.69) | 14.17 (18.65)

10. Secondary Outcome: Pre-dose Plasma Concentration (Ctrough) of Pirfenidone at Week 20
Description: Pirfenidone pre-dose plasma concentration (Ctrough) at Week 20 was reported applying the exclusion rules (e.g. dose reduction, discontinuation, samples flagged).
Time Frame: Week 20 (pre-dose)
Population: Participants in the PK analysis set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | GLPG1205 100 mg | Placebo
Number analyzed (Participants) | 4 | 6
ng/mL | 3701.0 (3583.1) | 2313.0 (1957.0)

ADVERSE EVENTS:
Time Frame: First dose date up to 30 days after the last dose of study drug (maximum up to 263 days)
Description: Full analysis set (FAS) consisted of all randomized participants who received at least 1 dose of study drug.
Arm/Group | GLPG1205 100 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 1/45 | 0/23
Serious Adverse Events (participants affected / at risk) | 9/45 | 1/23
Other Adverse Events (participants affected / at risk) | 36/45 | 18/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GLPG1205 100 mg (N=45) | Placebo (N=23)
Bronchitis (Infections and infestations) | 0 | 1
Gastrointestinal viral infection (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GLPG1205 100 mg (N=45) | Placebo (N=23)
Diarrhoea (Gastrointestinal disorders) | 12 | 3
Nausea (Gastrointestinal disorders) | 13 | 2
Abdominal pain (Gastrointestinal disorders) | 5 | 0
Vomiting (Gastrointestinal disorders) | 4 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Chronic gastritis (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Mucous stools (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 6 | 4
Bronchitis (Infections and infestations) | 3 | 3
Diarrhoea infectious (Infections and infestations) | 1 | 0
Erythema migrans (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Gastrointestinal viral infection (Infections and infestations) | 1 | 0
Gingival abscess (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Oral fungal infection (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Tracheitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Headache (Nervous system disorders) | 11 | 4
Dizziness (Nervous system disorders) | 6 | 2
Burning sensation (Nervous system disorders) | 1 | 0
Dyskinesia (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Parkinson's disease (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthenia (General disorders) | 9 | 0
Fatigue (General disorders) | 6 | 0
Chest pain (General disorders) | 1 | 0
Hunger (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Thirst (General disorders) | 1 | 0
Weight decreased (Investigations) | 6 | 1
Alanine aminotransferase increased (Investigations) | 3 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 0
Gamma-glutamyltransferase increased (Investigations) | 3 | 0
Blood bilirubin increased (Investigations) | 2 | 0
Blood lactate dehydrogenase increased (Investigations) | 2 | 0
Blood pressure increased (Investigations) | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Brain natriuretic peptide increased (Investigations) | 1 | 0
Neutrophil count increased (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 5 | 0
Appetite disorder (Metabolism and nutrition disorders) | 1 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0
Irritability (Psychiatric disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 2 | 0
Neutrophilia (Blood and lymphatic system disorders) | 2 | 0
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Hypertension (Vascular disorders) | 3 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic mass (Hepatobiliary disorders) | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Polyuria (Renal and urinary disorders) | 2 | 0
Renal pain (Renal and urinary disorders) | 1 | 0
Diplopia (Eye disorders) | 1 | 0
Panophthalmitis (Eye disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Tooth extraction (Surgical and medical procedures) | 1 | 0

LIMITATIONS AND CAVEATS:
The study was not powered to detect statistical significance and was limited by its small sample size, high variability of the primary endpoint (FVC), and a high rate of early treatment discontinuations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must review and approve any results of the study or abstracts for professional meetings prepared by the investigator(s). Published data must not compromise the objectives of the study. Data from individual study centers in multicenter studies must not be published separately.

DOCUMENTS (2):
  • Study Protocol (2020-04-30): https://cdn.clinicaltrials.gov/large-docs/52/NCT03725852/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-04): https://cdn.clinicaltrials.gov/large-docs/52/NCT03725852/SAP_001.pdf